CLINICAL TRIAL: NCT03422042
Title: An Open-labeled, Randomized Controlled Trial Comparing Between Short Duration And Standard Fourteen Days Antibiotic Treatments In Patients With Acute Common Bile Duct Stone Cholangitis After Successful Endoscopic Biliary Drainage
Brief Title: Short Duration Versus Fourteen Days Antibiotic in Common Bile Duct Cholangitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 56-124-21-1-2
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2017-11

CONDITIONS: Acute Cholangitis; Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short duration of antibiotic (Active Comparator): group A: will received intravenous antibiotic until the temperature is less than 37.8 c for 72 hours, then antibiotic is discontinued
  Interventions: Other: Short duration of antibiotic
- Standard treatment of antibiotic (Active Comparator): group B: will received intravenous antibiotic for 7 days, and followed by oral antibiotic for 7 days, regardless of body temperature
  Interventions: Other: Standard treatment of antibiotic

INTERVENTIONS:
Other: Short duration of antibiotic — Patient will received intravenous antibiotic until the body temperature is less than 37.8 c fir 72, then antibiotic is discontinued.
  Other Names: G1
  Arms: Short duration of antibiotic
Other: Standard treatment of antibiotic — Patient will received intravenous antibiotic for 7 days, followed by oral antibiotic for 7 days, regardless of the body temperature.
  Other Names: G2
  Arms: Standard treatment of antibiotic

SUMMARY:
Common bile duct stone cholangitis is a potentially fatal condition, characterized by an obstruction and bacterial infection of biliary system. The principles of management are appropriate biliary drainage and systemic antibiotics. There has been limited data about appropriate time of antibiotics in patient with successful endoscopic drainage.

DETAILED DESCRIPTION:
The aim is comparing the efficacy and safety between short duration and standard fourteen days antibiotic treatment in patients with acute common bile duct stone (CBDS) cholangitis after successful endoscopic biliary drainage as regards recurrence rate of acute cholangitis, complete stone clearance rate, morbidity and mortality associated acute cholangitis, and complications related ERCP procedure.

The study will be divided patients with acute CBDS cholangitis with complete stone clearance into 2 groups, group (A) will be received intravenous antibiotic until the temperature is less than 37.8 c for 72 hours and group (B) will be received intravenous antibiotic for 7 days, followed by oral antibiotic for 7 days, regardless of the body temperature.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* diagnosis of acute mild to moderate severity of ascending common bile duct stone cholangitis
* endoscopic retrograde cholangiopancreatography (ERCP) with biliary drainage within 72 hours after admission

Exclusion Criteria:

* pregnant woman
* the cause of obstruction other than common bile duct stone
* severe co-morbid diseases such as cardiovascular/pulmonary/kidney disease
* active concomitant infections of other organs
* history of allergy to cephalosporin group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-13 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
The recurrence rate of cholangitis | 8 weeks
  The number of patients who has recurrence of fever after complete treatment without other sources identified

SECONDARY OUTCOMES:
The rate of adequacy of drainage | 24 hours
  The number of patient with cholangiography at the end of the procedure showed no fill defect in the bile duct.
Complication rate | 4 weeks
  The number of patients who developed complications related procedure included pancreatitis, bleeding, perforation, cholangitis as defined and graded according to the consensus guideline and sedation related complications.
Mortality rate | 4 weeks
  The number of patient with death

CONTACTS AND LOCATIONS:
Overall Officials: Nisa Netinatsunton, MD., Principal Investigator — NKC Institute of Gastroenterology and Hepatology.
Locations (1):
- NKC Institue of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
The individual data of patients participating in the study are not available for public sharing since the investigators did not obtain the consent to share the data of patient